CLINICAL TRIAL: NCT06990217
Title: Comparison of Oxytocin Dosing Regimen' Low Versus High, in Gravida Women With BMI 30 and Above Undergoing Induction of Labor
Brief Title: Comparing High Versus Low Dose of Oxytocin, in Gravida Women With BMI 30 and Above Which Are Undergoing Induction of Labor
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Rola Iskander, Dr Rula Iskander - ObGyn resident and official investigator, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0022-24-EMC
Record Dates: First submitted 2025-05-07; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Induction of Labor; Augmentation of Labor
Keywords: induction of labor; augmentation of labor; obese; obese gravida; high dose of oxytocin in obese gravida
MeSH Terms: conditions — Obesity | interventions — Solutions; Injections

STUDY DESIGN:
Intervention Model Description: the two study groups will get the same drug but different dosage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High dose oxytocin (Active Comparator): This arm of the study will receive high dose oxytocin - 20 units of oxytocin in 1000 ml STD. Starting rate 12 ml/h increase dose by 12 ml/h every 30 min up to 5 contractions / 10 min. Max dose 120 ml/h.
  Interventions: Drug: Oxytocin Grindeks 10 IU/ml- solution for injection
- Low dose oxytocin (Other): This arm of the study will receive low dose oxytocin- - 10 units of oxytocin in 1000 ml STD. Starting rate 12 ml/h increase dose by 12 ml/h every 30 min up to 5 contractions / 10 min. Max dose 120 ml/h.
  Interventions: Drug: Oxytocin Grindeks 10 IU/ml- solution for injection

INTERVENTIONS:
Drug: Oxytocin Grindeks 10 IU/ml- solution for injection — our study is aims to compare two oxytocin regimens - low VS high dose among obese women who need induction or augmentation of labor

SUMMARY:
The goal of this clinical trial is to compare between higher and lower dose of oxytocin to induce delivery in obese women. Researches will compare between low and high doses of oxytocin. the study group will use high dose of oxytocin (20 units in 1000 ml) versus the control group which will use low dose of oxytocin (10 units of oxytocin in 1000 ml)

DETAILED DESCRIPTION:
the duration and the progression of the first stage of labor is slower in obese women and oxytocin seems to be less effective in the treatment of protracted labor in obese women. There is no consensus in the literature about the optimal oxytocin dose. Hence, the objective of this study is to compare 2 oxytocin regimens, low VS high dose among obese women who need induction or augmentation of labor.

Women at term (37-42 weeks), requiring the use of oxytocin for induction of labor or for augmentation of labor. Who are obese (BMI 30 and above), Viable singleton pregnancies with Cephalic presentation. After their consent, will be randomization: in a 1:1 allocation.

Group 1 (control) will receive a low dose- 10 units of oxytocin in 1000 ml STD. Starting rate 12 ml/h increase dose by 12 ml/h every 30 min up to 5 contractions / 10 min. Max dose 120 ml/h.

Group 2 (study) will receive a high dose- 20 units of oxytocin in 1000 ml STD. Starting rate 12 ml/h increase dose by 12 ml/h every 30 min up to 5 contractions / 10 min. Max dose 120 ml/h.

The primary outcome of the study is the time from the start of oxytocin to delivery

Statistical analysis Mean time interval from initiation of augmentation/ induction with oxytocin until delivery was eight hours (±240 minutes), based on previous observation at the delivery ward. The aim of study is to demonstrate a difference of 2 hours between the 2 groups with an alpha of 0.05 and a power of 80%, a sample size of 64 women per group is required. The primary analysis will be performed on the groups as allocated, that is, by the intention to treat, including all women as randomized.

ELIGIBILITY:
Inclusion Criteria:

* Women at term (37-42 weeks), requiring the use of oxytocin for induction of labor or for augmentation of labor.
* BMI 30 and above
* Viable singleton pregnancies
* Cephalic presentation.
* No contraindication for vaginal delivery

Exclusion Criteria:

* Women with previous cesarean delivery
* Multiple pregnancy
* Multiple fetal malformations
* IUFD

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only female gravida
Enrollment: 130 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time from the start of oxytocin to delivery | from the start of induction till delivery
  our hypothesis that high dose of oxytocin shortens the time from the start of induction to delivery

SECONDARY OUTCOMES:
Maternal age | at enrollment
  maternal age at enrollment
mode of delivery | at delivery
intrapartum fever | during labor
uterine rupture | up to 6 weeks after delivery
perineal tears | during delivery
PPH | up to 6 weeks
length of postpartum stay | perinatal.
  normally a gravida's length of stay after normal delivery is 48 hours and after c-section is up to 3-4 days.
Maternal satisfaction | will be assessed up to 1 day after delivery
  We will assess maternal satisfaction using a scale - Birth Satisfaction Scale-Revised (BSS-R). a five pont scale, 0 is totally disagree, 5 totally agree.
Neonatal outcomes | up to 1 week
  NICU admittion
Neonatal outcomes | up to 1 week
  neonatal PH<7.1
Apgar score | at 1, 5 and 10 minutes
  minimum 0 and maximum 10. zero is bad outcome 10 is good outcome
GTPAL system | at enrollment
  GTPAL system assessed by questionnaire
maternal weight | at enrollment
  weight before pregnancy, weight at admission
maternal height | at enrollment
  height

CONTACTS AND LOCATIONS:
Overall Officials: Rula Iskander, MD, Study Chair — Emek Medical Center
Locations (1):
- Haemek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No
to protect patients privacy.